CLINICAL TRIAL: NCT07178288
Title: Assessment of Pressure Pain Threshold (PPT) and Conditioned Pain Modulation (CPM) After Effect in Patients With and Without Tennis Elbow (TE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hashemite University (Other)
Responsible Party: Principal Investigator, Ahmad Muhsen, Assistant Professor, The Hashemite University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 32/1/2024/2025
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Tennis Elbow; Health Adult Subjects; Lateral Elbow Tendinopathy (Tennis Elbow); Pressure Pain Threshold (PPT); Conditioned Pain Modulation (CPM)
Keywords: Lateral elbow tendinopathy (tennis elbow), pressure pain threshold (PPT), conditioned pain modulation (CPM)
MeSH Terms: conditions — Tennis Elbow; Ceroid lipofuscinosis, neuronal 1, infantile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PPT_CPM Arm (Experimental): Procedure After completing self reported questionnaires, participants will attend a single test session where they undergo a Pressure Pain Threshold (PPT) test-retest protocol followed by a Conditioned Pain Modulation (CPM) testing protocol, with a rest period of 10 minutes in between. The experimental protocols will be performed by the same investigator. All instructions will be standardized
  Interventions: Other: Physiological/measurement-validation study

INTERVENTIONS:
Other: Physiological/measurement-validation study — Protocols PPT Reliability The assessor measured Pressure Pain Threshold; PPT, using an electronic digital algometer. Measurements will be taken at two test sites wrist at baseline, at 1, 3 and 5 minutes. Three PPT measurements were taken at each time point with a 15-20 seconds interval between each. Mean values will then be used in analysis.
  Conditioned Pain Modulation In order to assess CPM, PPT was used as a tested stimulus on the painful arm (elbow and wrist). Baseline PPTs will assessed three times with an interval of 30 seconds between the repetitions. A Cold Pressure Task (CPT) will be used as the conditioning stimulus. Participants will be instructed to immerse their uninvolved hand in the ice water for 2 minutes. PPT will be measured at baseline pre and 1 minute during immersion to calculate CPM response, and then at various time points post immersion (minutes: 1, 5, 15, 30, 45, and 60) to determine the time point at which PPT returns to baseline.

SUMMARY:
This study at Hashemite University looks at how people with and without tennis elbow (AKA lateral elbow tendinopathy) feel pressure pain and how their bodies briefly "turn down" pain after a cold stimulus. Participants complete brief questionnaires (basic demographics without names, a tennis-elbow symptom form, and a physical-activity form) and then have their pressure-pain threshold (PPT) tested with a handheld device that slowly increases pressure on standard spots near the elbow and wrist; they say when it first becomes painful. To test the body's built-in anti-pain system (conditioned pain modulation, CPM), one hand is placed in ice water (the cold-pressor task) and PPT is measured again at set times (before, during, and after the cold stimulus) to see how much pain sensitivity changes and how long that change lasts. Both PPT reliability and CPM after effect are measured in this study. The study findings may help improve future assessment and treatment of musculoskeletal pain conditions.

DETAILED DESCRIPTION:
This is a quasi-experimental reliability and time-course study using digital algometry for PPT and the cold-pressor task for CPM. Primary outcomes include PPT reliability (with intraclass correlation coefficient (ICC), standard error of measurement (SEM), and smallest detectable change (SDC) and the duration of CPM after-effects (time to return toward baseline). Testing is planned in the Physiotherapy Clinic at the Community Rehabilitation Center, with a minimum sample noted in the application. The protocol emphasizes standardized sites, repeated measures at predefined time points, and storage of coded data on university systems.

ELIGIBILITY:
TE Group

Inclusion Criteria:

Patients with Tennis Elbow confirmed at initial assessment by the Primary Investigator (PI)

Unilateral elbow pain > 6 weeks duration reproduced on at least two of the following tests:

* Palpation of the lateral epicondyle
* Isometric testing of the wrist extensors
* Middle finger extension test
* Passive stretch of wrist extensors
* Resisted hand gripping using a dynamometer
* Upper limb neurodynamic test-radial nerve bias (ULNDT-RN)

Exclusion Criteria:

* History of chronic pain conditions (e.g. fibromyalgia, irritable bowel
* syndrome, temporomandibular dysfunction, migraines)
* Neurological or sensory dysfunction (especially in the upper limbs)
* History of chronic musculoskeletal pain (e.g. arthritis, chronic low back
* pain)
* Contraindications to cold application (i.e. Reynaud's disease, diabetes)
* Current or long-term use of pain medication or anti-depressants

Healthy Group The asymptomatic group included adults (18-65 years) without pain (acute or chronic) at least 3 months before the experimental sessions.

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) | The PPT session would take about 30min to be completed in one day.
  The assessor measured PPT (kPa) using an electronic digital algometer (Somedic AB, Sweden). Measurements will be taken at two test sites wrist at baseline, at 1 minute, at 3 minutes and at 5 minutes. Three PPT measurements were taken at each time point with a 15-20 seconds interval between each. Mean values will then be used in analysis.
  PPT: the amount of pressure (measured with a handheld algometer in kPa) at the moment pressure first becomes painful.
  Intra/inter-rater reliability of PPT: how consistent PPT readings are when the same/and another tester repeats the measurements (ICC, SEM)
Conditioned Pain Modulation (CPM) | 1 and half hours in a separate day (different to the PPT session day)
  In order to assess Conditioned Pain Modulation (CPM), Pressure Pain Threshold (PPT) is used as a tested stimulus on the painful arm (elbow and wrist). Baseline PPTs is assessed three times with an interval of 30 seconds between the repetitions. A Cold Pressure Task (CPT) is used as the conditioning stimulus. Participants is instructed to immerse their uninvolved hand in the ice water for 2 minutes. PPT is measured at baseline prior to CPT, after 1 minute during immersion (CPT) to calculate CPM response, and then at various time points post immersion (1 minute, 5 minutes, 15 minutes, 30 minutes, 45 minutes, and 60 minutes) to determine the time point at which PPT returned to the baseline value. At each time point, PPT is measured three times with 15 to 20 second rest intervals in between. The mean value of the three measurements at each time point is used for statistical analysis. CPM after-effect (when the CPM effect returns to the baseline value) is calculated in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Muhsen, Principal Investigator — The Hashemite University
Locations (1):
- The Hashemite University, Department of Physical Therapy; Community Rehabilitation Center Clinics, Zarqa, Zarqa Governorate, Jordan

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author upon reasonable request.
Supporting Information: SAP
Time Frame: Soon after the study published in a peer reviewed journal.
Access Criteria: Researchers interested in the field upon a resealable request from the PI, the dataset and/or the analyses will be shared.

REFERENCES:
- [Background] Oono Y, Nie H, Matos RL, Wang K, Arendt-Nielsen L. The inter- and intra-individual variance in descending pain modulation evoked by different conditioning stimuli in healthy men. Scand J Pain. 2011 Oct 1;2(4):162-169. doi: 10.1016/j.sjpain.2011.05.006. PMID 29913755
- [Background] Bilika P, Kalamatas-Mavrikas P, Vasilis N, Strimpakos N, Kapreli E. Reliability of Pressure Pain Threshold (PPT) and Conditioned Pain Modulation (CPM) in Participants with and without Chronic Shoulder Pain. Healthcare (Basel). 2024 Aug 31;12(17):1734. doi: 10.3390/healthcare12171734. PMID 39273758